CLINICAL TRIAL: NCT01503255
Title: A Stage 2 Cognitive-behavioral Trial: Reduce Alcohol First in Kenya Intervention
Acronym: RAFIKI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Moi University (Other); Syracuse University (Other); Indiana University (Other); Yale University (Other)
Responsible Party: Principal Investigator, Rebecca Papas, Assistant Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01AA020805 (NIH)
Record Dates: First submitted 2011-12-16; First posted 2012-01-04 (Estimated); Last update posted 2017-07-14 (Actual); Status verified 2017-07

CONDITIONS: Hazardous Drinking; Binge Drinking; HIV-infected
Keywords: CBT; alcohol; HIV; Kenya; paraprofessional
MeSH Terms: conditions — Binge Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cognitive behavioral group therapy (Experimental)
  Interventions: Behavioral: cognitive behavioral group therapy
- health education group (Active Comparator)
  Interventions: Behavioral: health education group

INTERVENTIONS:
Behavioral: cognitive behavioral group therapy — 6 weekly 90-minute group sessions
  Arms: cognitive behavioral group therapy
Behavioral: health education group — 6 weekly 90-minute group sessions
  Arms: health education group

SUMMARY:
This study will determine whether a group cognitive-behavioral therapy intervention that demonstrates preliminary evidence of reducing alcohol use among HIV-infected outpatients in western Kenya is effective when compared against a group health education intervention in a large sample over a longer period of time. It will be delivered by paraprofessionals, individuals with limited formal education and little or no relevant professional experience. This approach is consistent with successful cost-effective models of service delivery in resource-limited settings in which paraprofessionals (e.g., clinical officers, traditional birth attendants and peer counselors) are trained.

DETAILED DESCRIPTION:
Hazardous and binge drinking have been associated with increased risky sexual behavior, poor adherence to antiretroviral therapy (ARVs) and toxicity from ARVs among those with HIV infection. As such, hazardous and binge drinking (score of e3 on the Alcohol Use Disorders Test - Consumption (AUDIT-C), or e6 drinks per occasion at least monthly) have a major impact on HIV transmission and disease progression. Prevalence rates of hazardous drinking are particularly high among HIV (53%) and general medicine (68%) outpatients in western Kenya, in part due to the wide availability of potent traditional brew. Growing evidence suggests that heavy drinking is an obstacle to successful sexual risk reduction approaches. This team recently completed a Stage 1 trial of a group cognitive-behavioral therapy (CBT) intervention delivered by paraprofessionals to reduce alcohol use among 74 HIV-infected Kenyans (R21AA017884). Results demonstrated feasibility, acceptability and estimated a large treatment effect at post-treatment. Investigators now propose a large Stage 2 efficacy trial of the CBT alcohol intervention. The goal is to evaluate the efficacy of the Reduce Alcohol First in Kenya Intervention (RAFIKI) in its ability to reduce alcohol use within a larger Stage 2 trial that includes an active control and a longer follow-up period. Rafiki means friend in Kiswahili, the national language of Kenya. The trial will be conducted by the Kenya Health Behavior Study (KHBS) team, an experienced group of Kenyan and U.S. behavioral scientists, physicians, substance users in recovery and persons infected with HIV. KHBS expands on well-established ties between the Academic Model for Providing Access to Healthcare (AMPATH) and the Brown University Medical School, which has been an active AMPATH partner since 1997. AMPATH currently treats more than 75,000 HIV-infected patients in 25 clinics in western Kenya. As part of these efforts, investigators have ready locally adapted training, treatment and fidelity rating manuals, a successful paraprofessional intervention delivery model, clinical assessment tools, and an experienced local team of trainers and supervisors. The specific aims are to: 1) To examine the efficacy of a same-sex group CBT intervention in a randomized clinical trial of 336 HIV-infected Kenyan outpatients who report hazardous or binge drinking, when compared to a time-matched group Healthy Lifestyles education intervention; 2) To conduct analyses to examine the mechanisms of intervention effects; and 3) To conduct exploratory analyses to examine the relationship between intervention condition and sexual risk behaviors. Completion of these objectives, which are consistent with NIAAA's mission to reduce both alcohol use and HIV risk in vulnerable populations, will provide a robust test of efficacy of the paraprofessionally led group CBT and potentially provide a sustainable and transportable intervention for other settings in sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18
* HIV infected outpatient enrolled in 1 of 5 AMPATH clinics
* drank alcohol in past month
* hazardous or binge drinker (AUDIT-C)
* lives within an hour of Eldoret HIV clinic
* verbal working knowledge of Kiswahili

Exclusion Criteria:

* active psychosis, suicidality or severe cognitive impairment
* physically unable to attend session
* previous participation in CBT study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2012-07; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Timeline Followback alcohol use (percent drinking days) | longitudinal alcohol use from baseline (past 30 days) to 9 month post-intervention follow up
  The Timeline Followback is a well-established, reliable and valid retrospective calendar-based measure employing memory cues to assess alcohol use. The primary hypothesis is that CBT will be more effective than HL in reducing alcohol use (percent drinking days) from baseline (past 30 days) through the 6-week active treatment phase. The secondary hypothesis is that CBT will be more effective than HL in reducing alcohol use (percent drinking days) from baseline through the 9-month post-intervention follow-up. Results will be analyzed in a longitudinal model.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Papas, PhD, Principal Investigator — Brown University
Locations (1):
- Moi University, Eldoret, Kenya

REFERENCES:
- [Derived] Galarraga O, Gao B, Gakinya BN, Klein DA, Wamai RG, Sidle JE, Papas RK. Task-shifting alcohol interventions for HIV+ persons in Kenya: a cost-benefit analysis. BMC Health Serv Res. 2017 Mar 28;17(1):239. doi: 10.1186/s12913-017-2169-4. PMID 28351364